CLINICAL TRIAL: NCT00449735
Title: Quinolone Resistance in Bloodstream Isolates of Escherichia Coli
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO07030003
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Bacterial Infections
Keywords: positive isolates; ecoli; blood cultures; positive cultures for ecoli; blood stream infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This proposed study aims to document the risk factors for quinolone resistance in bloodstream isolates of E. coli. Additionally, the adequacy of empiric antibiotic therapy for E. coli bloodstream infections will be assessed. Finally, outcome will be recorded - this is all-cause mortality at 28 days from the time of the first positive blood culture. Hypothesis: Ciprofloxacin resistant strains are associated with admission from nursing home and with prior quinolone use.

DETAILED DESCRIPTION:
The following information will be collected: age, sex, occupation, hospital location at the time of positive culture (ER, medical ward, ICU etc), date of positive culture, prior hospitalization, receipt of outpatient dialysis, home care or other regular medical care (eg, outpatient chemotherapy), presence of invasive devices, receipt of antibiotics, including their type and whether they were adequate for the resistance profile of the organism, prior positive microbiologic cultures, time and location of positive cultures, underlying diseases and severity of illness, presence of urinary or intravascular devices, recent immunomodulative therapies or radiation therapy, physical exam findings, laboratory and radiographical data, antimicrobial usage within 30 days of onset of the infection, microbiological data and resistance patterns, choice of antibiotics once organism identified, bacteriological outcomes, laboratory results, demographic information, medications, clinical outcome,gender, height, weight, ethnicity, and past medical history. We will collect information retrospectively.

ELIGIBILITY:
Inclusion Criteria:

Clinical information is collected by chart review of "case" and "control" patients.

A "case A" patient is defined as follows:

* One or more blood cultures are positive for E. coli. The organism is ciprofloxacin resistant.

A "case B" patient is defined as follows:

* One or more blood cultures are positive for E. coli. The organism is ciprofloxacin susceptible. Additionally, 4 controls who are in hospital at the same time as cases will be selected for each case.

Exclusion Criteria:

* If they do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: E coli positive cultures
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
dead or alive | end of study
  health status

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States